CLINICAL TRIAL: NCT04644107
Title: Expanded Access for Marizomib
Status: No longer available | Type: Expanded Access
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: Marizomib
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Solid Tumor
Keywords: Expanded Access; Compassionate Use
MeSH Terms: interventions — marizomib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Marizomib — Marizomib will be administered via IV
  Other Names: CC-92763

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to Marizomib.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Myers Squibb, Summit, New Jersey, United States